CLINICAL TRIAL: NCT00751374
Title: Prospective, Randomized, Open-Label Study of Topical Antibiotic Prophylaxis at the Catheter Exit Site: Continuous Daily Gentamicin Cream Versus Cyclical Gentamicin Cream and Mupirocin 2% Cream Alternating at Monthly Basis.
Brief Title: Topical Gentamicin Cream Versus Alternating Gentamicin and Mupirocin Cream in Peritoneal Dialysis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kwong Wah Hospital (Other)
Collaborators: The Hong Kong Society of Nephrology (Other)
Responsible Party: Tong Mei Wa Gensy, Kwong Wah Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KW/FR/08-007
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Last update posted 2008-09-11 (Estimated); Status verified 2008-09

CONDITIONS: Rate of Exit Site Infection; Rate of Atypical Mycobacterial Infection; Rate of Peritoneal Dialysis
MeSH Terms: interventions — Gentamicins; Mupirocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group A (Other): Topical gentamicin cream
  Interventions: Drug: gentamicin
- Group B (Active Comparator): topical gentamicin cream alternates with mupirocin cream at monthly basis
  Interventions: Drug: gentamicin cream alternating with mupirocin cream

INTERVENTIONS:
Drug: gentamicin — topical gentamicin cream on daily basis
  Arms: group A
Drug: gentamicin cream alternating with mupirocin cream — topical gentamicin cream alternating with mupirocin cream at monthly basis
  Other Names: Gentamicin and mupirocin
  Arms: Group B

SUMMARY:
Catheter-related infection, namely exit site infection and peritonitis, is the commonest complication of peritoneal dialysis. This complication causes significant morbidity and mortality in patients requiring peritoneal dialysis. Topical application of mupirocin 2% cream was first proven to be effective in reduction of staphylococcus-related catheter infection in 1990s. Subsequent randomized trial published in 2005 showed that gentamicin cream was superior to mupirocin 2% cream in reducing both Gram's positive and Gram's negative related catheter infection. However, a retrospective report published in 2007 puts the use of prophylactic antibiotic cream into a question. It reported an emergency of non-tuberculous mycobacterial infection in a dialysis center in Hong Kong after practising prophylactic application of gentamicin cream at the catheter exit site. The following prospective, randomized and open-label study aims to find out an optimal regimen of topical antibiotic prophylaxis in patients requiring peritoneal dialysis.

DETAILED DESCRIPTION:
Topical antibiotics therapy is a well-recognized prophylactic therapy towards the catheter exit site infection in peritoneal dialysis patient. Previous data has shown the superiority of gentamicin cream over the mupirocin cream in this aspect. However, the efficacy of the combination therapy using gentamicin cream alternating with mupirocin cream has not been tested. There is a potention benefit of reducing drug resistant strain in the combination group theoretically.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged 18 years old or above
2. Patient has Tenckhoff catheter inserted
3. Patient is expected to continue his or her dialysis in our center in the subsequent 3 years

Exclusion Criteria:

1. Patient fails to sign the written consent
2. Patient known to have allergy to either gentamicin or mupirocin
3. Patient has suffered from peritonitis or exit site infection 30 days before the enrollment.
4. Patient, suffering from terminal illness, has life-expectancy of less than one year
5. Patient expected to undergo peritoneal dialysis for less than one year, such as patients planning for elective renal transplantation or suffering from acute renal failure necessitating dialysis while waiting for the kidney to recover.
6. Pregnant patient
7. Patient known to be non-compliant
8. Patient bound by another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2008-09; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Rate of Exit site infection | every 3 months

SECONDARY OUTCOMES:
Rate of peritonitis | every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Gensy MW Tong, MBChB, Principal Investigator — Kwong Wah Hospital
Locations (1):
- Kwong Wah Hospital, Hong Kong, Hong Kong